CLINICAL TRIAL: NCT02507076
Title: Isolated Limb Perfusion for Advanced Melanoma or Sarcoma Limited to Extremity With or Without Distant Metastases
Brief Title: Isolated Limb Perfusion With Melphalan in Treating Patients With Stage IIIB-IV Melanoma or Sarcoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no enrollment
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-12-411; NCI-2013-01218 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-103; 11-12-411 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Basal Cell Carcinoma of the Skin; Eccrine Carcinoma of the Skin; Recurrent Adult Soft Tissue Sarcoma; Recurrent Melanoma; Recurrent Skin Cancer; Squamous Cell Carcinoma of the Skin; Stage III Adult Soft Tissue Sarcoma; Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Adult Soft Tissue Sarcoma; Stage IV Melanoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Sarcoma; Melanoma; Skin Neoplasms | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ILP with melphalan) (Experimental): Patients undergo ILP with melphalan IV over 60 minutes.
  Interventions: Drug: isolated limb perfusion; Drug: melphalan; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: isolated limb perfusion — Undergo ILP with melphalan
  Other Names: isolated limb infusion
Drug: melphalan — Undergo ILP with melphalan
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This pilot clinical trial studies isolated limb perfusion with melphalan in treating patients with stage IIIB-IV melanoma or sarcoma. Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Heating a chemotherapy solution and infusing it directly into the arteries around the tumor may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. This prospective trial will evaluate total response rate, including complete and partial response, in patients with unresectable extremity melanoma (or other skin cancer including but not limited to Merkel cell carcinoma) or soft tissue sarcoma treated with hyperthermic-isolated limb perfusion (ILP) with melphalan.

SECONDARY OBJECTIVES:

I. To evaluate the technical parameters including achievement of regional hyperthermia, arterial blood gas (ABG), tourniquet time, and their association with tumor response.

II. To evaluate time to recurrence and progression free survival (PFS) for patients with advanced extremity melanoma or sarcoma who achieved complete response after treatment with ILP with melphalan.

III. To evaluate overall survival rate and duration of survival for patients with advanced melanoma or sarcoma limited to extremity undergoing ILP with melphalan.

IV. To assess quality of life (QOL) score for patients undergoing ILP with melphalan.

OUTLINE:

Patients undergo ILP with melphalan intravenously (IV) over 60 minutes.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 4 months for 1 year, and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* The patient must have histological-proven primary or recurrent extremity melanoma (or other skin cancer including but not limited to Merkel cell carcinoma) or sarcoma, stage IIIB, IIIC, or IV (American Joint Committee on Cancer [AJCC] staging must be documented in patient's medical record, as determined by computed tomography [CT] of the chest, abdomen and pelvis, and/or whole body positron emission tomography [PET] scan, within six weeks prior to administration of study drug)
* Patients with stage IV disease who have high tumor burden and extensive symptomatic extremity disease
* Patients with stage IIIC disease must either have had regional lymph nodes previously removed or will have them removed either at the time of regional treatment or soon thereafter
* Disease to be treated by ILP must be unresectable and distal to the planned site of tourniquet placement (which for the leg is generally the apex of the femoral triangle, or for the arm is distal to the deltoid insertion)
* Patient's disease must be bi-dimensionally measurable by caliper or radiological method as defined in the Response Evaluation Criteria in Solid Tumors (RECIST) criteria (RECIST updated version 1.1); lesional tissue not necessary for diagnostic or other clinical purposes may be designated prospectively for research tissue banking
* Hemoglobin >= 8.0 g/dl
* White blood count (WBC) of >= 2000 m^3
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x the ULN
* Creatinine =< 1.5 x ULN
* Patient must have a palpable femoral/radial pulse in the affected extremity
* Patients must have a life expectancy of > 6 months
* Patient or the patient's legally acceptable representative must provide a signed and dated written informed consent prior to registration and any study-related procedures
* Patient or the patient's legally acceptable representative must provide written authorization to allow the use and disclosure of their protected health information at any institution subject to United States Health Insurance Portability and Accountability Act (US HIPAA) regulations; NOTE: This may be obtained in either the study-specific informed consent or in a separate authorization form and must be obtained from the patient prior to study registration

Exclusion Criteria:

* Cardiac disease: congestive heart failure > class II New York Heart Association (NYHA); patients must not have unstable angina (angina symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* Known brain metastasis; patients with neurological symptoms must undergo a CT scan/magnetic resonance imaging (MRI) of the brain to exclude brain metastasis
* Known human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Active clinically serious infection > Common Terminology Criteria for Adverse Events (CTCAE) grade 2
* Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event >= CTCAE grade 2 within 4 weeks of ILP/isolated limb infusion (ILI); any other hemorrhage/bleeding event >= CTCAE grade 3 within 4 weeks ILP/ILI
* Major surgery or significant traumatic injury within 30 days of ILI/ILP
* Evidence or history of bleeding diathesis or coagulopathy
* Antineoplastic therapy, radiotherapy, or any other investigational drug within 30 days prior to first study drug administration
* Patients with symptoms or signs of vascular insufficiency; specifically, patients with any history of blood clots or lifestyle altering ischemic peripheral vascular disease will be excluded
* History of allergic reactions and/or hypersensitivity to melphalan
* Psychiatric conditions or diminished capacity that could compromise the giving of informed consent, or interfere with study compliance
* Pregnant or nursing women are not eligible for this study
* Unable to return at the regular required intervals for reassessment, or study drug administration
* Patients with known heparin induced thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete and partial response) assessed by the RECIST v1.1 | Up to 12 weeks
  Rates of complete and partial response will be computed and reported with their 95% confidence intervals.

SECONDARY OUTCOMES:
Time to recurrence | Up to 4 years
  Kaplan-Meier methods will be used. 95% confidence intervals will be computed using Greenwood's formula.
Progression-free survival | Time of ILP procedure to date of recurrence, assessed up to 4 years
  Kaplan-Meier methods will be used. 95% confidence intervals will be computed using Greenwood's formula.
Overall survival | Time of ILP treatment to time of death, assessed up to 4 years
  Kaplan-Meier methods will be used. 95% confidence intervals will be computed using Greenwood's formula.

CONTACTS AND LOCATIONS:
Overall Officials: Katia Papalezova, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States